CLINICAL TRIAL: NCT04140058
Title: Hemodynamic Protection of Preoperative Ondansetron 15 Minutes Before Spinal Anaesthesia in Caesarean Section, a Prospective, Randomized Double Blind Study
Brief Title: Hemodynamic Protection of Preoperative Ondansetron 15 Minutes Before Spinal Anaesthesia in Caesarean Section
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Subhi M. Alghanem, Prof. of Anesthesia and Intensive care, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2433/2016/10
Record Dates: First submitted 2019-10-13; First posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Hypotension; Nausea; Vomiting
Keywords: Ondansetron; hypotension; nausea and vomiting; cesarean section
MeSH Terms: conditions — Hypotension; Nausea; Vomiting | interventions — Ondansetron; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group O4 (Active Comparator): Patients received 4mg ondansetron.
  Interventions: Drug: Ondansetron
- group O6 (Active Comparator): Patients received 6mg ondansetron.
  Interventions: Drug: Ondansetron
- group C (Placebo Comparator): Patients received normal saline.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ondansetron — ondansetron was administered 20 minutes prior to spinal anesthesia.
  Arms: group O4; group O6
Drug: Normal saline — Placebo of 10 mL normal saline was administered.
  Arms: group C

SUMMARY:
Spinal anaesthesia for caesarean section is the most commonly used anaesthetic choice in caesarean deliveries. This is usually associated with maternal hypotension and other adverse side effects. Prophylactic intravenous administration of ondansetron immediately and 5 minutes preoperatively have shown to provide a protective effect against hypotension while other studies have shown little effect on the incidence of blood pressure drop in healthy parturients.

The investigators will study the effect of different doses and timing of intravenous ondansetron in full term obstetric patients undergoing elective lower segment caesarean section under spinal anaesthesia on the incidence and severity of hypotension and other adverse side effects in healthy parturients having the standard intrathecal plain bupivacaine and fentanyl.

DETAILED DESCRIPTION:
This prospective randomized double-blind placebo-controlled study will include 150 American Society of Anaesthesiologist physical status grade I (ASA I) pregnant women scheduled for elective caesarean delivery under spinal anaesthesia.

Patients will be randomly allocated into three groups (n = 50) to receive intravenous ondansetron 4mg in 10 mL normal saline (group O4), 6 mg in 10 mL normal saline(group O6), or placebo of 10 mL normal saline (group C), all 15-20 minutes before spinal anaesthesia.

Hemodynamic variables and other adverse effects will be assessed at 16 time points intraoperatively. Those variables include blood pressure, heart rate, oxygen saturation, nausea, vomiting, electrocardiographic changes, skin flushing, discomfort or pruritus, perioperative vasopressor requirements and patients' satisfaction.

Participants will be randomly allocated preoperatively as per randomizer.org software and will be blinded from other anaesthetists performing the spinal block and following patients intraoperatively.

ELIGIBILITY:
Inclusion Criteria:

* patients who received spinal anesthesia for elective cesarean sections and meet the American Society of Anesthesiologist's (ASA) patient status classification I or II.

Exclusion Criteria:

* Patients ASA patient status classification III, IV or V
* Emergent cesarean sections
* Multiple parities (twins/triplets)
* More than 1,000 ml blood loss
* More than 6 mg ondansetron administered
* Patients presenting with a cardiac history (coronary artery disease, myocardial infarction, congestive heart failure, murmur, mitral valve prolapse/regurgitation, dysrhythmias, aortic stenosis/regurgitation)
* Patients presenting with preeclampsia
* Patients presenting for cesarean section with epidural due to failure to progress.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — full-term pregnant females undergoing cesarean section.
Enrollment: 151 (Actual)
Dates: Start 2016-01-02 (Actual); Primary Completion 2017-01-02 (Actual); Study Completion 2017-01-02 (Actual)

PRIMARY OUTCOMES:
Usage of Ondansetron prophylactically to prevent a significant decrease in systolic, diastolic, and mean blood pressure after the induction of spinal anaesthesia. | 1 year
  Baseline values of Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP), and Mean Blood Pressure (MBP) were recorded. Ondansetron was given 15 minutes before induction of spinal anesthesia. After initiation of spinal anesthesia, the SBP, DBP, and MBP were recorded regularly until the end of the cesarean section by a blinded anaesthesiologist.

SECONDARY OUTCOMES:
Prevention of intraoperative nausea and vomiting. | 1 year
  Patients were assessed for nausea, and vomiting throughout the whole intraoperative period by asking and observing the patients for any signs and/or symptoms of nausea, and we recorded any incident of intraoperative vomiting using the following scale:
  0) no any complaint.
  1. mild degree of nausea.
  2. moderate degree of nausea and vomit.
  3. frequently vomit.
  4. severely (continuously vomit.

CONTACTS AND LOCATIONS:
Locations (1):
- Jordan University Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No
No identifying information will be collected. Data will be used solely for statistical analysis.